CLINICAL TRIAL: NCT07128043
Title: The Effect of Cassava Waxes Hot Bath on Pain, Pressure Pain Threshold and Hand Function Among Patient With Trigger Finger: Single-Blind Randomized Controlled Trial Study
Brief Title: The Effect of Cassava Waxes Hot Bath on Pain, Pressure Pain Threshold and Hand Function Among Patients With Trigger Finger
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Phayao (Other)
Responsible Party: Principal Investigator, Chonticha Kaewjoho, Department of Physical Therapy, School of Allied Health Sciences, University of Phayao
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NarongsakMFU2568
Record Dates: First submitted 2025-07-31; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Patients With Trigger Finger
MeSH Terms: interventions — Ultrasonic Therapy

STUDY DESIGN:
Intervention Model Description: Arm 1:
  Name: Cassava waxes hot bath group ( Experimental group)
  Type: Experimental
  Description: Ultrasound therapy combined with cassava wax hot immersion
  Arm 2:
  Name: Control or comparison group
  Type: Active Comparator (Control)
  Description: Ultrasound therapy only
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound therapy combined with cassava wax hot immersion (Experimental): ultrasound therapy combined with cassava wax hot immersion group and ultrasound therapy only
  Interventions: Device: ultrasound therapy and cassava wax hot immersion
- ultrasound therapy (Sham Comparator): ultrasound therapy
  Interventions: Device: ultrasound therapy

INTERVENTIONS:
Device: ultrasound therapy and cassava wax hot immersion — participants sat in a comfortable position with their hand placed on a pillow or cushion. Ultrasound gel was applied to the base of the painful finger, and ultrasound therapy was performed for 5 minutes at a frequency of 3 MHz and an intensity of 0.5-1 W/cm. Afterward, the hand was cleaned and immersed in cassava wax heated to 125°F (51.7°C). The affected hand was dipped into the wax for 3 seconds, then removed. This process was repeated for 10 cycles. The hand was then wrapped in a plastic bag and a towel for 15 minutes before the wax was removed and peeled off.
  Arms: ultrasound therapy combined with cassava wax hot immersion
Device: ultrasound therapy — 1. ultrasound therapy Ultrasound gel was applied to the base of the painful finger, and ultrasound therapy was performed for 5 minutes at a frequency of 3 MHz and an intensity of 0.5-1 W/cm.
  Arms: ultrasound therapy

SUMMARY:
Objective: This study aimed to evaluate the efficacy of cassava wax hand immersion combined with ultrasound therapy on pain severity, pain threshold, finger locking frequency, and hand functional ability in patients with trigger finger. We assessed immediate, short-term, and long-term treatment outcomes.

Methods: This was a randomized controlled trial. Thirty-eight eligible volunteers were randomly assigned to two groups. The experimental group received ultrasound therapy combined with cassava wax hand immersion, while the control group received ultrasound therapy alone. Treatments were administered three times per week for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of trigger finger by a physician or a specialized physical therapist
* Present with all of the following symptoms: pain at the base of the affected finger, triggering (catching/locking) as a primary symptom (though pain often increased with it), and a palpable or audible triggering sensation during finger flexion and extension.
* Able to understand and follow the research procedures.

Exclusion Criteria:

* Having a history of neurological conditions, such as stroke or diseases causing sensory impairment in the upper limbs.
* Having arthritis or infection in the upper limbs
* Having Rheumatoid Arthritis.
* Having a skin condition in the wrist or hand area, upper limb fractures within the last 6 months, or those affecting movement.
* Having musculoskeletal deformities of the upper limbs that impact movement.
* Having an inflammation (e.g., pain, swelling, redness, warmth) in the wrist and fingers
* Having a history of upper limb surgery, an allergy to cassava starch/flour.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | - Time 1: Baseline or Day 1 - Time 2:After treatment, the first time of immediate effect - Time 3: After treatments in 4 weeks - Time 4: 1 month after finishing treatments in 4 weeks.
  This assesses the current pain severity using a 10-centimeter scale. Scores range from 0 to 10, where the far left end of the scale indicates "no pain at all" (score of 0), and the far right end indicates "worst pain imaginable" (score of 10). Participants were asked to mark an 'X' on the scale at the point corresponding to their current pain severity.
Pressure pain threshold | - Time 1: Baseline or Day 1 - Time 2:After treatment, the first time of immediate effect - Time 3: After treatments in 4 weeks - Time 4: 1 month after finishing treatments in 4 weeks.
  Participants were seated, and the assessor identified the location of the myofascial trigger point. This spot was marked with a washable pen. An algometer (a device used to measure pain threshold) was then applied to the marked trigger point at a rate of approximately 1 kg/second. Participants were instructed to signal immediately upon feeling the onset of pain (pain threshold). The applied pressure ranged from 0 to 11 kg/cm. Each participant underwent three measurements, with a 3-minute rest interval between each. The average of these three measurements was then calculated.
Pain frequency | - Time 1: Baseline or Day 1 - Time 2: After treatments in 4 weeks - Time 3: 1 month after finishing treatments in 4 weeks.
  Participants were interviewed regarding the frequency of finger locking symptoms and the number of finger locking episodes per day.
Disability of the arm, shoulder and hand | - Time 1: Baseline or Day 1 - Time 2: After treatments in 4 weeks - Time 3: 1 month after finishing treatments in 4 weeks.
  This is a questionnaire designed to assess the level of upper extremity impairment. It evaluates the functional ability of the wrist and finger joints, comprising 30 questions related to the patient's daily life activities and work capacity.

CONTACTS AND LOCATIONS:
Locations (1):
- Narongsak Khamnon, Chiang Rai, Tha Sut, Thailand

IPD SHARING:
Plan to Share IPD: No